CLINICAL TRIAL: NCT04594564
Title: Squeaking in Ceramic-on-Ceramic Total Hip Arthroplasty Using Delta TT Cup
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: LIMA Korea (Unknown)
Responsible Party: Principal Investigator, Young-Kyun Lee, Professor, Seoul National University Hospital
Other Study IDs: Delta TT cup
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis, Hip; Osteonecrosis of Femoral Head; Femoral Neck Fractures; Rheumatoid Arthritis of Hip; Posttraumatic Arthropathy
Keywords: Total hip arhtroplasty; Squeaking; Dislocation; Ceramic bearings
MeSH Terms: conditions — Osteoarthritis, Hip; Femur Head Necrosis; Femoral Neck Fractures; Joint Dislocations | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Total hip arthroplasty with Delta TT cup — Total hip arthroplasty using Delta TT cup and ceramic bearings

SUMMARY:
This study will evaluate clinical outcome on patients who undergo ceramic on ceramic (CoC) bearing total hip arthroplasty (THA) using Delta TT cup.

DETAILED DESCRIPTION:
This study will evaluate clinical outcome on patients who undergo ceramic on ceramic (CoC) bearing total hip arthroplasty (THA) using Delta TT cup. Specifically the study intends to address the following research topics:

1. The incidence of squeaking after CoC THA using Delta TT cup.
2. The dislocation rate and survival rate of CoC THA using Delta TT cup.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Non-inflammatory degenerative joint disease such as osteoarthritis or avascular necrosis
* Rheumatoid arthritis
* Post-traumatic arthritis
* Fractures of femoral neck

Exclusion Criteria:

* Local or systemic infection
* Septicaemia
* Persistent acute or chronic osteomyelitis
* Confirmed nerve or muscle lesion compromising hip joint function
* Unstable medical illness
* Rapidly progressive neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who undergo THA for their advanced hip disease.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Squeaking | 6 weeks
  Rate of any noise after THA
Squeaking | 3 months
  Rate of any noise after THA
Squeaking | 6 months
  Rate of any noise after THA
Squeaking | 9 months
  Rate of any noise after THA
Squeaking | 12 months
  Rate of any noise after THA
Squeaking | 24 months
  Rate of any noise after THA

SECONDARY OUTCOMES:
Dislocation | 6 weeks
  Dislocation rate after THA
Dislocation | 3 months
  Dislocation rate after THA
Dislocation | 6 months
  Dislocation rate after THA
Dislocation | 9 months
  Dislocation rate after THA
Dislocation | 12 months
  Dislocation rate after THA
Dislocation | 24 months
  Dislocation rate after THA

OTHER OUTCOMES:
Range of motion | 24 months
  Change of range of motion after THA
Survivorship of implant | 24 months
  Survival rate of prosthesis

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kyun Lee, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No